CLINICAL TRIAL: NCT03694574
Title: Emotion Regulation in Individuals With High and Low Trait Schizotypy. A Randomized Controlled Trial Comparing Suppression and Reappraisal
Brief Title: Emotion Regulation in Trait Schizotypy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danube University Krems (Other)
Collaborators: University of Vienna (Other)
Responsible Party: Principal Investigator, Krisztina Kocsis-Bogar, academic staff, Danube University Krems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DanubeUK
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Trait Schizotypy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low schizotypy (Other): Schizotypy score < 14 measured by the German Version of Schizotypal Personality Questionnaire (Klein, Andresen, & Jahn, 1997)
  Interventions: Behavioral: instruction to suppress; Behavioral: instruction to reappraise; Behavioral: control
- High schizotypy (Other): Schizotypy score ≥ 14 measured by the German Version of Schizotypal Personality Questionnaire (Klein, Andresen, & Jahn, 1997)
  Interventions: Behavioral: instruction to suppress; Behavioral: instruction to reappraise; Behavioral: control

INTERVENTIONS:
Behavioral: instruction to suppress — "It might happen that in some situations in which you try to do something and you fail or things don't come up as you want, you could become angry, mad or irritated and feel some level of distress and discomfort. Next, try not to think of the situation that makes you angry, mad or irritated. Please try as much as you cannot to think about the situation, don't think about how you feel or what had happened, and try to suppress your emotions and not to feel them. It's very important to try as much as you cannot to think about the situation that makes you angry, mad or irritated." (Szasz, Szentagothai, & Hoffmann, 2011)
Behavioral: instruction to reappraise — "It might happen that in some situations in which you try to do something and you fail or things don't come up as you want, you could become angry, mad or irritated and feel some level of distress and discomfort. Next, please try to tell yourself that or would be preferable that the others are nice and/or fair to you, but if they are not, it does not mean that you or they are worthless human beings. It would be preferable that the others be nice and/or fair to you but if they are not, remember that it is only (very) bad), not catastrophic (the worst thing that could happen to you). It would be preferable that others are nice and/or fair to you, but if they are not, you can tolerate it, and go on enjoying life, even if it's more difficult at the beginning." (Szasz et al., 2011)
Behavioral: control — No instruction

SUMMARY:
Our aim is to compare state anger and state emotion regulation strategies in healthy individuals with high trait schizotypy and to look at differences of induced anger, negative emotions, decrease of positive emotions and aggressive behaviour after anger induction. Our further aim is to compare conditions where an instruction to suppress or reappraise emotions is given with a control condition with no instruction.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 58 years,
* good command of German language

Exclusion Criteria:

* present or past psychiatric or neurological illness,
* ongoing treatment with psychiatric drugs,
* constant consume of heroin or hallucinogenic drugs,
* alcohol dependence,
* cannabis consume two weeks before testing.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
state anger | 3 minutes
  measured by the German version of State-Trait Anger Expression Inventory (Schwenkmetzger, Hodapp, & Spielberger, 1992)
state negative emotions | 3 minutes
  measured by the German Version of Positive and Negative Affect Schedule (Krohne, Egloff, Kohlmann, & Tausch, 1996)
state positive emotions | 3 minutes
  measured by the German Version of Positive and Negative Affect Schedule (Krohne, Egloff, Kohlmann, & Tausch, 1996)
aggressive behavior | 3 minutes
  measured by the amount of chili measured by the Hot Sauce Paradigm (Lieberman, Solomon, Greenberg, & McGregor, 1999)

IPD SHARING:
Plan to Share IPD: Undecided
Interested researchers can request the data from the primary investigator (krisztina.kocsis-bogar@donau-uni.ac.at). Please give a short description of the study including an explanation about how you are going to use the data.

REFERENCES:
- [Background] Klein, C., Andresen, B., & Jahn, T. (1997). Erfassung der schizotypen Persönlichkeit nach DSM-III-R: Psychometrische Eigenschaften einer autorisierten deutschsprachigen Übersetzung des
- [Background] Krohne, H. W., Egloff, B., Kohlmann, C. W., & Tausch, A. (1996). Untersuchung mit einer deutschen Form der Positive and Negative Affect Schedule (PANAS). Diagnostica, 42, 139-156.
- [Background] Lieberman, J. D., Solomon, S., Greenberg, J. & McGregor, H. A. (1999). A hot new way to measure aggression: hot sauce allocation, Aggressive Behavior, 25, 331-348
- [Background] Schwenkmetzger, P., Hodapp, V., & Spielberger, C. D. (1992). Das State-Trait-Ärgerausdrucks-Inventar (STAXI). Bern: Huber.
- [Background] Szasz PL, Szentagotai A, Hofmann SG. The effect of emotion regulation strategies on anger. Behav Res Ther. 2011 Feb;49(2):114-9. doi: 10.1016/j.brat.2010.11.011. Epub 2010 Dec 9. PMID 21185551